CLINICAL TRIAL: NCT01703364
Title: Fludarabine/Rituximab Combined With Escalating Doses of Lenalidomide in Untreated Chronic Lymphocytic Leukemia (CLL) - a Dose-finding Study With Escalating Starting Dose of Lenalidomide and Concomitant Evaluation of Safety and Efficacy
Brief Title: Fludarabine/Rituximab Combined With Escalating Doses of Lenalidomide in Untreated CLL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_CLL-9; 2011-004912-43 (EudraCT Number)
Record Dates: First submitted 2012-10-04; First posted 2012-10-10 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: CLL; Chronic Lymphocytic Leukemia
Keywords: CLL; Lenalidomide; Revlimid; AGMT; T cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide/Fludarabine/Rituximab (Experimental): Lenalidomide: day 8-21 of cycle 1 and day 1-21 of cycles 2-6; Starting Dose: 5 mg (first 5 patients) and 10 mg (further 5 patients) increase Lenalidomide dose via dose levels (10)/15/20/25 mg/d every 28 days if no limiting toxicity occurs
  Fludarabine: 25 mg/m2 iv d1-3 or 40 mg/m2 po d1-3; repeat every 28 days
  Rituximab: 375 mg/m2 iv day 4 on cycle 1 and 500 mg/m2 iv day 1 on cycles 2-6; repeat every 28 days
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide: day 8-21 of cycle 1 and day 1-21 of cycles 2-6; Starting Dose: 5 mg (first 5 patients) and 10 mg (further 5 patients) increase Lenalidomide dose via dose levels (10)/15/20/25 mg/d every 28 days if no limiting toxicity occurs
  Fludarabine: 25 mg/m2 iv d1-3 or 40 mg/m2 po d1-3; repeat every 28 days
  Rituximab: 375 mg/m2 iv day 4 on cycle 1 and 500 mg/m2 iv day 1 on cycles 2-6; repeat every 28 days
  Other Names: Revlimid

SUMMARY:
This is a trial in patients with previously untreated CLL. Eligible patients will receive Lenalidomide with a backbone of Fludarabine and Rituximab for 6 therapy cycles. Lenalidomide will be increased by dose steps of 5 mg every cycle in the absence of limiting toxicity. If limiting toxicity ensues the patients will be treated with last tolerable dose for the remainder of the 6 treatment cycles.

The first 5 patients will start with dose level 5 mg Lenalidomide and further escalating dose. After the fifth patient is included in the study, enrolment will be interrupted until this patient has finished his first treatment cycle. A safety board will evaluate the toxicities of the first 5 patients. If there are more than 2 patients experiencing a dose limiting toxicity (DLT) in the first treatment cycle, the starting dose will not be escalated and further 5 patients will be enrolled with a starting dose of 5 mg Lenalidomide. If only 2 or less patients experience a DLT in the first treatment cycle, the next 5 patients will start the treatment with 10 mg Lenalidomide.

The rational for the higher starting doses stems from the lack of tumor lysis or tumor flare toxicity in this combination on the one hand and from the observation that the very slow escalation from 2,5 mg on led to a lack of efficacy in monotherapy trials due to early progression in a relevant number of cases. The increase of the Lenalidomide dosage should result in an increased efficacy especially at the beginning and a higher cumulative dose of Lenalidomide.

The identification of patients intolerant to Lenalidomide by immunophenotyping of the T cells for validation is also part of this trial, because intolerance seems to be not dose dependent but may be caused by T cell activation. Therefore, early identification of patients intolerant to this form of modern immunochemotherapy and establishing efficient Lenalidomide based combination therapy is an important part of improvement of current CLL treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female ≥ 18 years of age
* CLL (as determined by CD23+, CD5+, CD19+)
* Treatment indication as defined by the NCI Workshop criteria (see appendix 6 and reference 10)
* ECOG ≤ 2
* No previous treatment of the CLL by chemotherapy, radiotherapy (except localized radiotherapy of 1 lymphatic area) or immunotherapy
* Life expectancy > 6 months (except prognosis due to high risk CLL)

Exclusion Criteria:

* Active bacterial, viral or fungal infection
* Positivity for HIV, Hepatitis B or C
* Patients with known history of thromboembolic events
* Reduced organ functions and bone marrow dysfunction not due to CLL
* Creatinine clearance of below 30 ml/min
* Patients with known history of thromboembolic events
* Patients with a history of other malignancies within 2 years prior to study entry (except for adequately treated carcinoma in situ of the cervix; basal or squamous cell skin cancer; low grade, early stage localized prostate cancer treated surgically with curative intent; good prognosis DCIS of the breast treated with lumpectomy alone with curative intent)
* Patients with medical co-morbid conditions that would require long term use (> 1 month) of systemic corticosteroids during study treatment
* Patients with a history of severe cardiac disease; e.g. NYHA Functional Class III or IV heart failure, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, or unstable angina
* Other known co-morbidity with the potential to dominate survival
* Transformation to aggressive B-cell malignancy (e.g., large B-cell lymphoma, Richter's syndrome, or prolymphocytic leukemia (PLL))
* Hypersensitivity with anaphylactic reaction to humanised monoclonal antibodies or any of the applied drugs
* Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol
* Administration of any investigational agent(s) within 4 weeks prior to entry
* Pregnancy or lactation
* Medical or psychological condition which in the opinion of the Investigator would not permit the patient to complete the study or sign meaningful informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-06; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Tolerability of escalated starting dose | 12 month, 20 month
  Interim analysis after completion of cylce 1 of the first 5 patients, final analysis after last pastient last visit Metrics: Number of patients experiencing defined dose limiting toxicities during cycle 1

SECONDARY OUTCOMES:
Establishment of maximal tolerated dose (MTD) of Lenalidomide in combination with FR | 20 month
Time to MTD | 20 month
Safety profile of the FRL combination | 20 month
  Analysis of occuring adverse events during the study treatment according to Common Terminology Criteria for Adverse Events (CTCAE)
Response rates in all phases by 4-colour flow cytometric and ASO-PCR MRD analysis | 20 month
Risk factor analysis (FISH cytogenetics, CD38/ZAP-70 expression, mutation status) | 20 month
Longitudinal definition of T cell subsets (including prognostic EM T cells and Treg cells)+/- PD1 | 20 month

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Universitätsklinik der PMU Salzburg, Univ-Klinik für Innere Medizin III, Salzburg, Salzburg
  - Universitätsklinik für Innere Medizin Innsbruck, Klinische Abteilung für Hämatologie und Onkologie, Innsbruck, Tyrol

REFERENCES:
- See also: AGMT — http://www.agmt.at